CLINICAL TRIAL: NCT01427010
Title: A Feasibility Study on Adaptive 18F-FDG-guided Radiotherapy for Recurrent and Second Primary Head and Neck Cancer in the Previously Irradiated Territory.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011/536
Record Dates: First submitted 2011-08-29; First posted 2011-09-01 (Estimated); Last update posted 2018-04-19 (Actual); Status verified 2018-04

CONDITIONS: Re-irradiation in Recurrent and Second Primary Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Intervention Model Description: Feasibility study
Oversight: Data Monitoring Committee: No

ARMS (1):
- Reirradiation of recurrent and 2nd primary head/neck cancer. (Experimental)
  Interventions: Radiation: [18F]FDG-PET-voxel intensity-based IMRT

INTERVENTIONS:
Radiation: [18F]FDG-PET-voxel intensity-based IMRT — Non-controlled, non-randomized, prospective study on 18F-Fluorodeoxyglucose-Positron Emission Tomography ([18F]FDG-PET)-voxel intensity-based intensity-modulated radiotherapy (IMRT) (dose painting) adapted to the anatomical and biological changes as detected by per-treatment FDG-PET/Computertomography (CT) acquired at the end of the 2nd and the 4th week of treatment.

SUMMARY:
Adaptive dose painting appears to increase the chance of cure at minimized radiation-induced toxicity in intensity-modulated radiotherapy (IMRT) for primary head and neck cancer. This could also be of importance in IMRT for recurrent and second primary head and neck cancers in previously irradiated territory.

This trial investigates the feasibility of continuous adaptive 18F-Fluorodeoxyglucose-Positron Emission Tomography-voxel ([18F]FDG-PET-voxel) intensity-based IMRT in reirradiation of patients with recurrent and second primary head and neck cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed recurrences and second primary squamous cell carcinoma of the oral cavity, oropharynx, hypopharynx or larynx in the previously irradiated territory.
* Primary unresectable tumor and/or patients refused surgery.
* No grade 3 or more late toxicity (except xerostomia) after the initial radio(chemo)therapy for primary head and neck cancer.
* Minimal interval 12 months after the initial radio(chemo)therapy for primary head and neck cancer.
* Decision of a multidisciplinary tumor board on curative radiotherapy (in combination or not with targeted therapy with cetuximab)
* Karnofsky performance status ≥70%.
* Age ≥ 18 years old.
* Informed consent obtained, signed and dated before specific protocol procedures.

Exclusion Criteria:

* Previous radiotherapy for cT1-2 cN0 M0 glottic cancer.
* Brachytherapy as treatment for second primary / recurrence.
* Distant metastases.
* Other second primary tumors that are not under control.
* Pregnant or lactating women.
* Elevated blood creatinine level.
* Allergy to the CT-contrast agents.
* Mental condition rendering the patient unable to understand the nature, scope, and possible consequences of the study.
* Patient unlikely to comply with protocol, i.e. uncooperative attitude, inability to return for follow-up visits, and unlikely to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
To test success rate of continuous adaptive 18F-Fluorodeoxyglucose-Positron Emission Tomography ([18F]FDG-PET)-guided radiotherapy (intensity-modulated radiotherapy (IMRT) and/or helical tomotherapy). | 2 year
  To test feasibility of continuous adaptive 18F-Fluorodeoxyglucose-Positron Emission Tomography ([18F]FDG-PET)-guided radiotherapy (intensity-modulated radiotherapy (IMRT) and/or helical tomotherapy) in treatment of recurrent and second primary head and neck cancer in the previously irradiated territory.

SECONDARY OUTCOMES:
Estimation time to progression. | At 6, 9 and 12 months
Evaluation tumor response. | After 3 months.
Number of Participants with Adverse Events. | Up to 3 months.
  Evaluation acute toxicity.

CONTACTS AND LOCATIONS:
Overall Officials: Wilfried De Neve, Ph.D., M.D., Principal Investigator — University Hospital, Ghent
Locations (2):
- Belgium (2):
  - Antwerp University Hospital, Antwerp
  - University Hospital Ghent, Ghent

REFERENCES:
- See also: Related Info — http://www.uzgent.be